CLINICAL TRIAL: NCT00280163
Title: Genomics and Postoperative Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lawrence Wei, Associate Professor, University of Pittsburgh
Other Study IDs: 0506010
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Atrial Fibrillation, Genomics
Keywords: Genomics, cardiac surgery

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

SUMMARY:
This research study is done to find out if genetic make up of a person plays a role in complications and recovery after the Coronary Artery Bypass Graft (CABG) operation.

As you may be aware, the DNA (Deoxyribonucleic acid) is a chemical in our body that carries the genetic information. There are common but very small variations (polymorphisms) that occur in DNA. We would like to find out if these common variations put a person at increased risk for developing complications- especially rapid irregular heart beat after the CABG operation.

DETAILED DESCRIPTION:
Postoperative Atrial Fibrillation has been shown to increase the length of hospital stay; markedly increase cost and potentially increases the incidence of post-operative stroke. Nationally, postoperative atrial fibrillation (AF) is a common complication of cardiac surgery, occurring in 25% to 40% of patients and total costs of billions of dollars per year to treat At University of Pittsburgh Presbyterian University Hospital, over the past few years, our patients experience AF in the postoperative period at an average rate of 30% -40%. The incidence of postoperative AF increases with the age of the patient. The average age of the patient that undergoes CABG surgery has been on the increase due to the improved longevity of the population.

Coronary artery bypass grafting is associated with systemic inflammatory response. There have been studies performed to assess the relationship of genetic polymorphisms that could affect the expression of cytokines such as interleukin 6 (IL-6). Interleukin 6 is a pro-inflammatory cytokine and major mediator of acute phase response. The correlation between the -174 G/C polymorphism and the high production of IL-6 has enabled some investigators to anticipate and treat the patients prophylactically to reduce the IL-6 levels. 8

It has been suggested that inflammation can have a role in the development of atrial arrhythmias after cardiac surgery and that genetic predisposition to develop postoperative complications exists. There have been studies performed in Europe to ascertain this association and it has been found that the -174G/C Interleukin-6 promoter gene variant appears to modulate the inflammatory response to surgery and to influence the development of postoperative AF. These data suggest an inflammatory component of postoperative atrial arrhythmias and a genetic predisposition to this complication , this polymorphism has also been correlated with the development of postoperative renal and pulmonary complications.

Enrolled patients will have a single blood sample of 6 ml drawn prior to their CABG surgery.

Any personal identifiers on the blood sample tube will be removed and code numbers specific for this research study will be affixed on to the samples by the research coordinator before the samples are sent to the Genomics laboratory for analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are about to have a Coronary Artery Bypass Grafting Surgery done.

Exclusion Criteria:

* Inability or unwilling to provide an informed consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients about to undergo or have undergone Coronary Artery Bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2005-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Wei, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC PUH, Pittsburgh, Pennsylvania, United States